CLINICAL TRIAL: NCT04052464
Title: The Study of the Implantation Window From Endometrial Biopsy With Gene Expression Methods
Status: Completed | Type: Observational
Sponsor: Prelife Kft (Industry)
Responsible Party: Principal Investigator, Balint Laszlo Balint, Principal Investigator, Prelife Kft
Other Study IDs: PRELIFE-V8
Record Dates: First submitted 2019-08-06; First posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Infertility, Female; IVF
Keywords: gene expression; biomarkers; implantation window; embryo transfer; endometrium; biopsy; lavage; liquid biopsy
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- endometrium biopsy only: In these cases, only endometrium biopsy is investigated for the selected biomarkers gene expression profile.
  Interventions: Other: endometrium biopsy
- endometrium lavage followed by endometrium tissue biopsy: In these cases before the endometrium tissue biopsy, an endometrial lavage is performed and from both samples, the selected biomarkers gene expression profile are investigated.
  Interventions: Other: endometrium biopsy; Other: endometrium lavage
- serial endometrium lavage followed by endometrium biopsy: In these cases before the endometrium tissue biopsy, at different days endometrial lavage samples are taken. From all samples, the selected biomarkers gene expression profile are investigated.
  Interventions: Other: endometrium biopsy; Other: repeated endometrium lavage

INTERVENTIONS:
Other: endometrium biopsy — All patients will have endometrium biopsy.
Other: endometrium lavage — In some selected cases biopsy is preceded by endometrium lavage.
  Groups: endometrium lavage followed by endometrium tissue biopsy
Other: repeated endometrium lavage — Endometrium lavage is repeated during the same cycle.
  Groups: serial endometrium lavage followed by endometrium biopsy

SUMMARY:
The objective of the study is to gain a better understanding of the gene expression changes in the endometrial biopsy especially whether the endometrium has reached a receptive status, i.e. the implantation window, or not.

DETAILED DESCRIPTION:
The endometrium goes through huge gene expression changes during a cycle, the cells are transformed, the mucous membrane thickens, then loosens, and finally sheds. In this process, the expression of the genes also goes through significant changes, which can be determined from a small tissue sample.

Endometrium biopsy samples can be used for endometrium phasing. A question of the study is the feasibility of using for endometrium phasing beside endometrium tissue biopsy also samples generated by endometrium lavage. The advantage of this latter method is that it is minimally invasive, it does not cause haemorrhage and has minimal side effects. In some selected cases endometrial lavage will be performed on the same day with endometrial tissue sampling together with the drawing of a peripheral blood sample.

A list of potential biomarkers was proposed from the meta-analysis of published gene expression datasets. From the endometrium derived samples, RNA will be isolated and gene expression biomarkers will be measured. Expression profiles will be compared to published reference samples.

ELIGIBILITY:
Inclusion Criteria:

* infertile women participating in the diagnostic evaluation of infertility.

Exclusion Criteria:

* patients who are legally incapable or partially capable
* pregnancy should be excluded before sampling
* bleeding problems
* the active phase of severe psychiatric disorders

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study aims to better understand the component of female infertility, therefore, is investigating only women.
Study Population: Infertile women participating in the diagnostic evaluation of infertility. The patients are contacted for participation in the study during the diagnostic evaluation of their infertility at specialized infertility or gynaecological clinic.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
gene expression profile | measurements are performed within 3 weeks after samples are shipped to the laboratory
  the endometrium derived samples are measured for the mRNA level expression of a selected list of biomarkers as it follows: ABCC3, ACTB, ADAMTS2, ADAMTS8, ARG2, ASPN, B2M, BAMBI, C10orf10, C1QTNF6, C2CD4A, CCDC71L, CD55, CEBPD, CP, CRISP3, CTHRC1, CYP24A1, CSRP2, DDX52, DPP4, DUOX1, DUOXA1, EDNRB, FCER1G, G0S2, GADD45G, GNG2, GNG4, GPX3, GRAMD1C, GREM2, GZMA, HPGD, HTR2B, IGFBP1, IGFBP3, IGFBP6, IL1B, IRX3, ITGA2, ITGB6, KAL1, KCND2, KCNK3, LCP2, LEFTY2, LRP4, LTBP2, LUM, MAOA, MAP2K6, MFSD4, MMP10, MS4A7, MT1M, MUC16, NID2, NNMT, OPRK1, PAEP, PDE4B, PHLDB2, PKHD1L1, PLAT, PLD1, POLR2A, PPIA, RARRES1, RDH10, RGS1, RHOB, RHPN2, RIMKLB, SGIP1, SLAIN1, SLC15A1, SLC15A2, SLC1A1, SLC26A7, SLC5A3, SOD2, SPP1, SYT11, TBP, TCN1, TFPI2, THBS1, TIMP3, TMC5, TMED6, TNFRSF11B, TSPAN8
endometrium phase assesment | phase assignment is performed within two weeks after the measurements are performed.
  based on the gene expression profile endometrium samples are phase assigned based on published reference samples

CONTACTS AND LOCATIONS:
Overall Officials: Balint L. Balint, MD, PhD, Principal Investigator — Prelife Kft

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared as the approval does not allow sharing of the individual participant data.